CLINICAL TRIAL: NCT06117787
Title: Blood Pressure Monitor#Model#KD-7920#Clinical Test
Brief Title: Blood Pressure Monitor Clinical Test (Cuff Range: 13.5cm-19.5cm）
Status: Completed | Type: Observational
Sponsor: Andon Health Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: Andon Health 13
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Blood Pressure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subject use both KD-7920 Wrist Automatic Electronic BPM and mercury sphygmomanometers

SUMMARY:
The purpose of this study is to verify the accuracy of the blood pressure cuffs with blood pressure monitor device.

Cuff circumference is 13.5cm-19.5cm.

ELIGIBILITY:
Inclusion Criteria:

* Normal blood pressure and hypertensive patients over 12 years old.

Exclusion Criteria:

* Patients with serious arrhythmias or a high frequency of arrhythmias
* Pregnant woman
* Other investigators believe that it is not suitable to participate in this clinical trial

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Normal blood pressure and hypertensive patients over 12 years old.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2022-04-02 (Actual); Primary Completion 2023-05-28 (Actual); Study Completion 2023-05-28 (Actual)

PRIMARY OUTCOMES:
blood pressure monitor accuracy | 30 minutes
  All the test results of the electronic blood pressure monitor with the cuff is within the accuracy creteria, with the merury sphygmomanometer as control

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, China